CLINICAL TRIAL: NCT01106482
Title: A Phase IV, Open-label, Multi-center Follow-up Study to Determine the Persistence of Tick-borne Encephalitis (TBE)-Specific Antibody Responses Among Children and Adolescents Previously Immunized Against TBE
Brief Title: An Extension Study to Determine the Persistence of Tick-borne Encephalitis (TBE)-Specific Antibody Responses Among Children and Adolescents Previously Immunized Against TBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M48P3E1
Record Dates: First submitted 2010-04-12; First posted 2010-04-20 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Tick Borne Encephalitis (TBE)
Keywords: TBE; Tick Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

ARMS (4):
- Arm 1 (Active Comparator)
  Interventions: Other: Serology blood draw
- Arm 2 (Active Comparator)
  Interventions: Other: Serology blood draw
- Arm 3 (Active Comparator)
  Interventions: Other: Serology blood draw
- Arm 4 (Active Comparator)
  Interventions: Other: Serology blood draw

INTERVENTIONS:
Other: Serology blood draw — Blood draw only, no vaccine

SUMMARY:
This study will evaluate the durability of antibody responses in children and adolescents after primary immunization with TBE vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy study subjects from the parent study who completed the primary vaccination series, with parental or legal guardian informed consent

Exclusion Criteria:

* Subjects who did not receive complete schedule of primary vaccination in the parent study
* Subjects enrolled in other investigational studies at the same time and within the last three months
* Subjects with any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Analysis of immunogenicity (TBE neutralizing antibody levels) 3 years after vaccination | 3 years after vaccination
Analysis of immunogenicity (TBE neutralizing antibody levels) 4 years after vaccination | 4 years after vaccination
Analysis of immunogenicity (TBE neutralizing antibody levels) 5 years after vaccination | 5 years after vaccination

SECONDARY OUTCOMES:
Analysis of immunogenicity (TBE antibody levels as measured by ELISA) at 3 years after vaccination | 3 years after vaccination
Analysis of immunogenicity (TBE antibody levels as measured by ELISA) at 4 years after vaccination | 4 years after vaccination
Analysis of immunogenicity (TBE antibody levels as measured by ELISA) at 5 years after vaccination | 5 years after vaccination

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - Winkelhoferstr. 3, Ehingen
  - Fuggerplatz 1, Kaufering
  - Hauptstrasse 240, Kehl
  - Bismarckstr. 3, Ludwigsburg
  - Am Marktplatz 8, Oberkirch
  - Großbottwarer Str. 47, Oberstenfeld
  - Wilhelmstr. 7, Offenburg
  - Stuttgarter Str. 74, Stuttgart
  - Martin-Niemöller-Str. 2, Traunreut
  - Murnauer Str. 3, Weilheim

REFERENCES:
- [Derived] Wittermann C, Izu A, Petri E, Gniel D, Fragapane E. Five year follow-up after primary vaccination against tick-borne encephalitis in children. Vaccine. 2015 Apr 8;33(15):1824-9. doi: 10.1016/j.vaccine.2015.02.038. Epub 2015 Feb 26. PMID 25728316